CLINICAL TRIAL: NCT03539328
Title: MITO27: Randomized Phase II Study on MK-3475 Plus Chemotherapy Versus Chemotherapy Alone in Recurrent, Platinum-resistant Ovarian Cancer
Brief Title: Study on MK-3475 Plus Chemotherapy Versus Chemotherapy Alone in Recurrent, Platinum-resistant Ovarian Cancer
Acronym: MITO27
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180-17
Record Dates: First submitted 2018-03-23; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; Gemcitabine; Paclitaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Other): Pegylated Liposomal Doxorubicin 40 mg/mq iv q 28 or Weekly Paclitaxel 80 mg/mq d 1,8,15 q 28 or Gemcitabine 1000 mg/mq d 1,8 q 21 or At physician' discretion
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel; Drug: Liposomal Doxorubicin
- Pembrolizumab (Experimental): Pegylated Liposomal Doxorubicin 40 mg/mq iv q 28 or Weekly Paclitaxel 80 mg/mq d 1,8,15 q 28 or Gemcitabine 1000 mg/mq d 1,8 q 21 or At physician' discretion plus Pembrolizumab 200 mg d1 q 21 iv infusion in 30 minutes
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Liposomal Doxorubicin

INTERVENTIONS:
Drug: Pembrolizumab — Humanized antibody used in cancer immunotherapy.
  Arms: Pembrolizumab
Drug: Gemcitabine — Chemotherapy medication
Drug: Paclitaxel — Chemotherapy medication
Drug: Liposomal Doxorubicin — Chemotherapy medication

SUMMARY:
The study is designed to assess the therapeutic efficacy and toxicity of the combination chemotherapy with pembrolizumab in recurrent, platinum resistant OC patients. The main objective is to test whether the therapeutic intervention benefits the patients evaluating the increase in overall survival with respect to chemotherapy alone.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label trial, designed to assess the therapeutic efficacy and toxicity of the combination chemotherapy with pembrolizumab in recurrent, platinum resistant OC patients. The main objective is to test whether the therapeutic intervention benefits the patients evaluating the increase in overall survival with respect to chemotherapy alone.

Eligible patients will be randomized 1:1 to receive:

ARM A:

Pegylated Liposomal Doxorubicin 40 mg/mq iv q 28 Weekly Paclitaxel 80 mg/mq d 1,8,15 q 28 Gemcitabine 1000 mg/mq d 1,8 q 21 At physician' discretion or

ARM B:

Pegylated Liposomal Doxorubicin 40 mg/mq iv q 28 Weekly Paclitaxel 80 mg/mq d 1,8,15 q 28 Gemcitabine 1000 mg/mq d 1,8 q 21 plus Pembrolizumab 200 mg d1 q 21 iv infusion in 30 minutes In both arms patients will receive treatments until disease progression, unacceptable toxicity of patient's refusal. Patients will receive at least 6 to 8 cycles of chemotherapy at physician's discretion. In the experimental arm patients who stop chemotherapy for toxicity reasons and whose disease is at least in stabilization, may continue treatment with Pembrolizumab as single agent.

Patients will be stratified according to the number of previous chemotherapy lines (1 vs >1) and measurable/evaluable disease.

ELIGIBILITY:
Inclusion Criteria:

1. Platinum resistant (platinum free interval 1-6 months from last platinum dose) ovarian, Fallopian tube or primary peritoneal cancer;
2. Be willing and able to provide written informed consent/assent for the trial;
3. Be 18 years of age on day of signing informed consent;
4. Have measurable disease or evaluable based on RECIST 1.1 (patients with only CA 125 increase without evidence of disease are not included);
5. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen;
6. Have a performance status of 0 or 1 on the ECOG Performance Scale;
7. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation;
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 6.5.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment;
2. Has received >2 previous CHT lines;
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment;
4. Has a known history of active TB (Bacillus Tuberculosis);
5. Hypersensitivity to pembrolizumab or any of its excipients;
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier;
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent:

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study;
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy;
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer and other solid tumors within the last 2 years;
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment;
11. Has an history of, or any actual evidence of active, non-infectious pneumonitis that required steroids treatment;
12. Has an active infection requiring systemic therapy;
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator;
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
15. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment;
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent;
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies);
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | from randomization to the date of death, assessed up to 44 months
  The combination of pembrolizumab and chemotherapy is expected to increase overall survival with respect to chemotherapy alone

SECONDARY OUTCOMES:
Progression free survival (PFS) | from randomization to the date of radiological/clinical progression of disease or death, assessed up to 44 months
  The combination of pembrolizumab and chemotherapy is expected to increase progression free survival with respect to chemotherapy alone
Response rate | 44 months
  The combination of pembrolizumab and chemotherapy is expected to increase response rate with respect to chemotherapy alone.
Adverse events | 44 months
  Incidence of adverse events, according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 5.0
Exploratory Objective: relationship between PD-L1 expression and response to Pembrolizumab treatment. | At screening phase: within 28 days before the start of treatment
  PD-L1 expression in tumor tissue will be characterized by immunohistochemistry to explore the relationship between tumor PD-L1 expression and response to treatment with pembrolizumab.
Exploratory Objective: association between anti-tumor activity from genetic alterations that may indicate a specific genotype reflective of greater dependency on PD-1/PD-L1 checkpoint function or other immune checkpoint signaling pathways | At screening phase (within 28 days before the start of treatment) and every 3 cycles (each cycle is 28 days), up to 44 months
  DNA isolated from blood or tumor tissue will be analyzed in order to identify genetic alterations and to evaluate specific genetic alterations that may correlate with clinical response to Pembrolizumab.
Quality of life | 44 months
  To assess patient-reported outcome (PRO) of patients receiving chemotherapy plus pembrolizumab with respect to patients receiving chemotherapy alone utilizing the disease-related symptoms - physical subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy FACT-Ovarian Symptom Index 18 (FOSI-18) Changes. The time to an event in PRO (Patient Reported Outcome) of worsening of disease symptoms will be defined as the time from randomization to a 4-point reduction in the FACT-O questionnaire.
Quality of life | 44 months
  To assess patient-reported outcome (PRO) of patients receiving chemotherapy plus pembrolizumab with respect to patients receiving chemotherapy alone using Euro- Quality of Life 5D tool, indicating which statements best describe the patient health state regarding: mobility, self-care, usual activities, pain/discomfort, anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Domenica Lorusso, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No